CLINICAL TRIAL: NCT03295110
Title: Lili Smart Study - Connected Solution of Assistance Dedicated to Caregivers and People With Alzheimer's Disease or Related Diseases
Brief Title: Connected Solution of Assistance Dedicated to Caregivers and People With Alzheimer's Disease or Related Diseases
Acronym: Lili smart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Lili smart (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 69HCL16_0706
Record Dates: First submitted 2017-09-12; First posted 2017-09-27 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease and Related Disorders (ADRD); natural caregiver; non-medical connected device; caregiver's burden; anxiety; costs; quality of life; depressive symptoms; independence
MeSH Terms: conditions — Alzheimer Disease; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functionalities of the Lili Smart Solution activated (Experimental): Lili Smart solution consists of an application for caregivers (web / mobile), a GSM watch worn by the patient, smart sensors placed at different locations of the patient's home and a support service 24 / 24 and 7/7.
  Interventions: Other: Functionalities of the Lili Smart Solution activated
- Functionalities of the Lili Smart Solution non activated (Other): Lili Smart watch worn by the participants and sensors placed at home with their functionalities inactivated. Absence of the web / mobile application.
  Interventions: Other: Functionalities of the Lili Smart Solution non activated

INTERVENTIONS:
Other: Functionalities of the Lili Smart Solution activated — Non-medical connected device (Lili Smart solution) activated : application for caregivers (web / mobile), GSM watch worn by the patient, smart sensors placed at different locations of the patient's home and a support service 24 /24 and 7/7.
  Other Names: Non-medical connected device (Lili Smart solution) with active functionalities
  Arms: Functionalities of the Lili Smart Solution activated
Other: Functionalities of the Lili Smart Solution non activated — Non-medical connected device (Lili Smart solution) with inactive functionalities : watch worn by the participants and sensors placed at home with their functionalities inactivated. Absence of the web / mobile application.
  Other Names: Non-medical connected device (Lili Smart solution) with inactive functionalities
  Arms: Functionalities of the Lili Smart Solution non activated

SUMMARY:
Alzheimer's disease and related diseases (ADRD) are a major public health issue. In France, nearly 900,000 people have ADRD, which represents about 70% of dementia cases, and the expected prevalence for 2020 is 1.2 million.

Patients with ADRD have cognitive, behavioral and functional impairments that lead to progressive impairment of quality of life and autonomy. Maintaining them at home depends predominantly on their caregivers, mainly family, spouse or child. By definition, the caregiver is "the person who provides partial or total support to an elderly dependent person or a person with a disability in the vicinity of the victim for the activities of daily life".

The investment of caregivers is therefore both human and financial, representing a greater or lesser burden. This burden can significantly affect their quality of life. Indeed, studies have shown that caregivers suffer from depletion, anxiety, depression and sleep disorders resulting in a deterioration of their health, leading them to greater care consumption. They would be more prone to cardiovascular diseases and cancer.

A review of the literature from 2009 examined 66 studies evaluating the contribution of various technologies targeting demented patients and their caregivers. Of these, only 10 dealt with independence at home and the well-being of the patient and his / her caregiver. The main limitations of these studies are the small samples (ranging from 1 to 6 patients), the degree of cognitive degradation (mainly moderately severe) and the lack of standardized assessment.

Although new technologies promise powerful home-based solutions, studies evaluating their efficacy for patients with ADRD and their caregivers remain scarce and fragile at the level of evidence due to methodological biases.

DETAILED DESCRIPTION:
Description of the intervention: Lili Smart solution consists of an application for caregivers (web / mobile), a GSM watch worn by the patient, smart sensors placed at different locations of the patient's home and a support service 24 / 24 and 7/7.

Objectives: The main objective is to evaluate the impact of the Lili Smart solution on the burden felt by caregivers of patients with ADRD at 3 months and at 6 months of follow-up.

The secondary objectives are to evaluate the impact of the Lili Smart solution at 3 months and 6 months of follow-up on:

* The anxiety of the caregiver of the patient with ADRD;
* Depression of the caregiver of the patient with ADRD;
* The quality of life of the caregiver of the patient with ADRD;
* The quality of life of the patient with ADRD,
* The level of functional autonomy of the patient with ADRD.
* The risks associated with the functional decline (falls, run aways) of the patient with ADRD.

In addition to the social impact measurement, the study aims to demonstrate the medico-economic impact of Lili smart solution as follow:

* The direct and indirect medical costs of the patient and the caregiver.

Patient and caregiver adherence to the Lili Smart solution will also be assessed as a secondary objective.

Methodology : This study is an interventional research on the human person meeting the definition 1 ° of article L1121-1 of the CSP and not relating to the products mentioned in article L. 5311-1 It is a randomized, controlled, single-blind, parallel-group, interventional, randomized, controlled trial in N = 60 patients and their primary caregiver with an observational phase (inactive device), and one interventional phase (activated device).

ELIGIBILITY:
Inclusion Criteria:

Caregiver inclusion's criteria :

* Natural caregiver helping the patient at least 6h / week for activities of daily living (if more than one caregiver, only one "referent" caregiver will be involved);
* Can be the caregiver of only one patient of the study.
* Having the ability to follow the study at the discretion of the investigator;
* Having agreed to participate in the study;
* Affiliated to a social security scheme;

Patient Inclusion Criteria:

* Diagnosis of Alzheimer's disease or related disease;
* Living at home
* Age ≥ 50 years
* Mini Mental State Examination (MMSE): 16-24 (included) (light to moderate);
* Affiliated to a social security scheme;
* Having agreed to participate in the study;
* Having the physical and psychic abilities to follow the study according to the appreciation of the investigator.

Exclusion Criteria:

Patients exclusion's criteria:

* Known psychiatric disorders
* Disabling motor and / or sensory impairment
* Patient under guardianship

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Caregiver's burden evolution | 6 months after randomization
  Natural caregiver's burden evolution after 6 months of follow-up. Natural caregiver's burden evolution after 6 months of follow-up. Assessement with the Zarit scale

SECONDARY OUTCOMES:
Evolution of the caregiver's anxiety level | 3 months and 6 months after randomization
  Evolution of the caregiver's anxiety level estimated with repeated measures with the Spielberger's State-Trait Anxiety Inventory (STAI Y-A / Y-B).
Evolution of the caregiver's depressive symptomatology | 3 months and 6 months after randomization
  Evolution of the caregiver's depressive symptomatology estimated with repeated measures of the Beck Depression Inventory (BDI)
Evolution of the caregiver's quality of life | 3 months and 6 months after randomization
  Evolution of the caregiver's quality of life estimated with repeated measures of the Quality of Life in Alzheilmer's Disease scale, caregiver version
Evolution of the patient's quality of life | 3 months and 6 months after randomization
  Evolution of patient's quality of life estimated with repeated measures of the Quality of Life in Alzheilmer's Disease scale, patient version
Evolution of the patient's independence | 3 months and 6 months after randomization
  Evolution of the patient's independence with repeated measures of the Instrumental Activities of Daily Life (IADL-E, 9 items).
Evolution of the caregiver's quality of life | 3 months and 6 months after randomization
  Evolution of the caregiver's quality of life estimated with repeated measures of the Quality of Life with EQ-5D questionnaire (EuroQol Five Dimensions questionnaire).
Evolution of the patient's quality of life | 3 months and 6 months after randomization
  Evolution of patient's quality of life estimated with repeated measures of the Quality of Life with EQ-5D questionnaire (EuroQol Five Dimensions questionnaire).
Number of falls | 1 months, 3 months and 6 months after randomization
  Number of times the patient has fallen after 1 month, 3 months and 6 months.
Number of run aways | 1 months, 3 months and 6 months after randomization
  Number of times the patient has ran away after 1 month, 3 months and 6 months.
Number of drugs prescribed to the caregiver and the patient | at inclusion and at 6 months
  Evolution of the number of drugs prescribed to the caregiver and the patient at inclusion and after 6 months of follow-up.
Indirect medical costs and direct non-medical costs | 6 months
  Data for indirect medical costs and direct non-medical costs will be collected with the RUD LITE questionnaire and the Lyon CMRR's MEMORA database
Evaluation of the caregiver's adherence to the Lili Smart solution | 7 months
  Evaluation of the caregiver's adherence to the Lili Smart solution after 7 months of follow-up (1 month of observation phase then 6 months of intervention) estimated through data collected in Lili Smart databases (number of connections to the application).
Evaluation of patient's adherence to the Lili Smart solution | 7 months
  Evaluation of the patient's adherence to the Lili Smart solution after 7 months of follow-up (1 month of observation phase then 6 months of intervention) estimated through data collected in Lili Smart databases (number of hours when the watch is worn).
Caregiver's burden evolution | 3 months after randomization
  Natural caregiver's burden evolution after 3 months of follow-up. Assessement with the Zarit scale

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak-Salmon, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital des Charpennes, Villeurbanne, France